CLINICAL TRIAL: NCT05372068
Title: Cement flooRs AnD chiLd hEalth (CRADLE): a Randomized Trial in Rural Bangladesh
Brief Title: Cement flooRs AnD chiLd hEalth (CRADLE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); North Carolina State University (Other); Soil Transmitted Helminthiasis Control Program, Directorate General of Health Services, Bangladesh (Unknown); Stanford Woods Institute for the Environment (Unknown)
Responsible Party: Principal Investigator, Jade Benjamin-Chung, Assistant Professor of Epidemiology & Population Health, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 63990; R01HD108196 (NIH)
Record Dates: First submitted 2022-05-06; First posted 2022-05-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Ascaris Lumbricoides Infection; Necator Americanus Infection; Trichuris Trichiura; Infection; Diarrhea
MeSH Terms: conditions — Trichuriasis; Diarrhea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concrete household floor (Experimental)
  Interventions: Other: Concrete household floor
- Non-intervention (No Intervention)

INTERVENTIONS:
Other: Concrete household floor — Household soil floors will be replaced with concrete floors
  Arms: Concrete household floor

SUMMARY:
This randomized trial in rural Bangladesh will measure whether installing concrete floors in households with soil floors reduces child enteric infection. The trial will randomize eligible households to receive concrete household floors or to no intervention and measure effects on child soil-transmitted helminth infection, diarrhea, and other enteric infections. The study will collect longitudinal follow-up measurements at birth and when children are ages 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Residence in Chauhali upazila or adjacent upazilas in Sirajganj or Tangail districts in Bangladesh
* No plan to relocate in the next 2-3 years
* Reside in home with floors made entirely of soil
* Pregnant woman 13-30 weeks gestation resides in the home at the time of enrollment

Exclusion Criteria:

* Home is not strictly residential (e.g., includes a business)
* Household with walls made of mud/soil
* Household floor size > 500 square feet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Child prevalence of any soil-transmitted helminth infection | Up to 24 months
  Prevalence of Ascaris lumbricoides, Necator americanus, or Trichuris trichiura infection in birth cohort detected with qPCR at 6, 12, 18, or 24 months follow-up

SECONDARY OUTCOMES:
Child Ascaris lumbricoides infection prevalence | Up to 24 months
  Prevalence of Ascaris lumbricoides infection in birth cohort detected with qPCR at 6, 12, 18, or 24 months follow-up
Child Necator americanus infection prevalence | Up to 24 months
  Prevalence of Necator americanus infection in birth cohort detected with qPCR at 6, 12, 18, or 24 months follow-up
Child Trichuris trichiura infection prevalence | Up to 24 months
  Prevalence of Trichuris trichiura infection in birth cohort detected with qPCR at 6, 12, 18, or 24 months follow-up
Child diarrhea prevalence | Up to 24 months
  Prevalence of diarrhea is defined as 3 or more loose or watery stools in 24 hours or 1 or more stools with blood in 24 hours at any follow-up measurement. Diarrhea will be based on caregiver-reported symptoms in the birth cohort with 2-day and 7-day recall at any follow-up measurement through month 24
Ascaris lumbricoides prevalence in household floor samples | Up to 24 months
  Prevalence of Ascaris lumbricoides in household floor dust detected with qPCR in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Necator americanus prevalence in household floor samples | Up to 24 months
  Prevalence of Necator americanus detected in household floor dust with qPCR in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Trichuris trichiura prevalence in household floor samples | Up to 24 months
  Prevalence of Trichuris trichiura detected in household floor dust with qPCR in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Any soil-transmitted helminth prevalence in household floor samples | Up to 24 months
  Prevalence of Ascaris lumbricoides, Necator americanus, or Trichuris trichiura detected in household floor dust with qPCR in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Culturable E. coli abundance in household floor samples | Up to 24 months
  Abundance (most probable number per square meter) of E. coli in household floor swabs detected with IDEXX in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Culturable E. coli abundance in child hand rinse samples | Up to 24 months
  Abundance (most probable number per two hands) of E. coli on child hands enumerated with IDEXX in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)
Culturable cefotaxime-resistant E. coli prevalence in household floor samples | Up to 24 months
  Prevalence of cefotaxime-resistant E. coli in household floor swabs detected with a modified IDEXX protocol with cefotaxime supplement in a sub-sample of households at any follow-up measurement (6, 12, 18, 24 months follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Jade Benjamin-Chung, PhD MPH, Principal Investigator — Stanford University
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All human subjects and environmental data will be de-identified and published. Identifiers that will be removed include participant names, address, date of birth, and geocoordinates. Coded data from videos will be made public, but videos will not be published in order to protect participant privacy. All data will be made available at the individual level (or household level, in the case of the household survey).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will be made publicly available within 2 years of the end of the study or at the time of publication, whichever is sooner.
Access Criteria: To be determined

REFERENCES:
- [Derived] Rahman M, Jahan F, Hanif S, Yeamin A, Shoab AK, Andrews JR, Lu Y, Billington S, Pilotte N, Shanta IS, Jubair M, Rahman M, Kabir M, Haque R, Tofail F, Hossain MS, Mahmud ZH, Ercumen A, Benjamin-Chung J. Effects of household concrete floors on maternal and child health: the CRADLE trial - a randomised controlled trial protocol. BMJ Open. 2025 Mar 3;15(3):e090703. doi: 10.1136/bmjopen-2024-090703. PMID 40032381
- [Derived] Rahman M, Jahan F, Hanif S, Yeamin A, Shoab AK, Andrews JR, Lu Y, Billington S, Pilotte N, Shanta IS, Jubair M, Rahman M, Kabir M, Haque R, Tofail F, Hossain S, Mahmud ZH, Ercumen A, Benjamin-Chung J. Effects of household concrete floors on maternal and child health - the CRADLE trial: a randomised controlled trial protocol. medRxiv [Preprint]. 2024 Jul 27:2024.07.26.24311076. doi: 10.1101/2024.07.26.24311076. PMID 39108529